CLINICAL TRIAL: NCT02587598
Title: A Phase 1/2 Study of INCB053914 in Subjects With Advanced Malignancies
Brief Title: Study of INCB053914 in Subjects With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 53914-101
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Solid Tumors
Keywords: leukemia; myelodysplastic syndrome (MDS); myelodysplastic/myeloproliferative neoplasms (MDS/MPN); myelofibrosis (MF); lymphoproliferative disorders; acute myeloid leukemia (AML); lymphomas; multiple myeloma (MM); PIM kinases
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders; Primary Myelofibrosis; Lymphoproliferative Disorders; Leukemia, Myeloid, Acute; Lymphoma; Multiple Myeloma | interventions — Azacitidine; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (9):
- Parts 1 and 2: INCB053914 100 mg QD (Experimental): INCB053914 will be self-administered orally once a day in as a 100mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914
- Parts 3 and 4: INCB053914 + Azacitidine (Experimental): Azacitidine will be administered at a dose of 75 mg/m2 subcutaneously or via IV per day, as a combination therapy with INCB053914.
  Interventions: Drug: INCB053914; Drug: Azacitidine
- Parts 3 and 4: INCB053914 + I-DAC (Intermediate dose cytarabine) (Experimental): I-DAC (intermediate dose cytarabine) will be administered at a dose of 1 g/m2 per day as an infusion as a combination therapy with INCB053914.
  Interventions: Drug: INCB053914; Drug: I-DAC (Intermediate dose cytarabine)
- Parts 3 and 4: INCB053914 + Ruxolitinib (Experimental): Ruxolitinib will be administered as an oral dose between 5 mg to 25 mg twice per day, as a combination therapy with INCB053914.
  Interventions: Drug: INCB053914; Drug: Ruxolitinib
- Parts 1 and 2: INCB053914 50 mg (Experimental): INCB053914 will be self-administered orally twice day in as a 50mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914
- Parts 1 and 2: INB053914 65 mg (Experimental): INCB053914 will be self-administered orally twice day in as a 65mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914
- Parts 1 and 2: INB053914 80 mg (Experimental): INCB053914 will be self-administered orally twice day in as a 80mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914
- Parts 1 and 2: INB053914 100 mg BID (Experimental): INCB053914 will be self-administered orally twice day in as a 100mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914
- Parts 1 and 2: INB053914 115 mg (Experimental): INCB053914 will be self-administered orally twice day in as a 115mg immediate release tablet as a monotherapy.
  Interventions: Drug: INCB053914

INTERVENTIONS:
Drug: INCB053914 — Initial cohort dose of INCB053914 at the protocol-specified starting dose in two treatment groups in dose escalation, with subsequent expansion in up to five cohorts based on protocol-specific criteria.
  INCB053914 tablets to be administered by mouth.
Drug: I-DAC (Intermediate dose cytarabine) — Cytarabine dose will be 1 g/m^2. Cytarabine will be administered as an intravenous (IV) infusion.
  Arms: Parts 3 and 4: INCB053914 + I-DAC (Intermediate dose cytarabine)
Drug: Azacitidine — Azacitidine dose will be 75 mg/m^2. Azacitidine will be administered either sub-cutaneously (SC) or intravenously (IV).
  Other Names: Vidaza®
  Arms: Parts 3 and 4: INCB053914 + Azacitidine
Drug: Ruxolitinib — Starting dose of ruxolitinib will be the dose the subject was on at study entry Ruxolitinib will be administered by mouth.
  Arms: Parts 3 and 4: INCB053914 + Ruxolitinib

SUMMARY:
This is an open-label, dose-escalation study of the proviral integration site of Moloney murine leukemia virus (PIM) kinase inhibitor INCB053914 in subjects with advanced malignancies. The study will be conducted in 4 parts. Part 1 (monotherapy dose escalation) will evaluate safety and determine the maximum tolerated dose of INCB053914 monotherapy and the recommended phase 2 dose(s) (a tolerated pharmacologically active dose that will be taken forward into the remaining parts of the study). Part 2 (monotherapy dose expansion) will further evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of the recommended Phase 2 dose(s). Part 3 (combination dose finding) will evaluate safety of INCB053914 in combination with select standard of care (SOC) agents and will identify the optimal INCB053914 dose in combination with conventional SOC regimens to take forward into Part 4. Part 4 (combination dose expansion) will further evaluate the safety, efficacy and pharmacokinetics of the recommended Phase 2 dose combination(s).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed diagnosis of select advanced malignancy
* Parts 1 and 2:

  * Unresponsive to currently available therapy and there is no standard-of-care therapy available in the judgment of the investigator.
  * Not currently a candidate for curative treatment
* Parts 3 and 4:

  * Subjects with relapsed/refractory AML must have received either induction chemotherapy for AML or hypomethylating agents for hematologic disease before AML.
  * Elderly subjects (≥ 65 years) with newly diagnosed AML must be treatment naive and unfit for intensive chemotherapy.
  * Myelofibrosis subjects must have been treated with ruxolitinib for ≥ 6 months with a stable dose for ≥ 8 weeks (acceptable doses are 5 mg twice daily [BID] to 25 mg BID).
* Willingness to undergo a pretreatment bone marrow biopsy and/or aspirate, or archival sample obtained since completion of most recent therapy (as appropriate to subjects with existing bone marrow disease or for whom bone marrow examination is a component of disease status assessment)
* Eastern Cooperative Oncology Group (ECOG) performance status

  * Part 1: 0 or 1
  * Parts 2, 3 and 4: 0, 1, or 2
* Life expectancy > 12 weeks or ≥ 24 weeks for Part 3 and Part 4 MF subjects.

Exclusion Criteria:

* Inadequate bone marrow or organ function
* Received an investigational agent within 5 half-lives or 14 days, whichever is longer, prior to receiving the first dose of study drug
* Received non-biologic anticancer medication within 5 half-lives prior to receiving the first dose of study drug (within 6 weeks for mitomycin-C or nitrosoureas), within 28 days for any antibodies or biological therapies
* Prior receipt of a PIM inhibitor
* Any history of disease involving the central nervous system (Part 1). Known active disease involving the central nervous system (Part 2).
* Screening corrected QT interval (QTc) interval > 470 milliseconds
* Radiotherapy within the 2 weeks prior to initiation of treatment
* Chronic or current active infection requiring systemic antibiotic, antifungal, or antiviral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, M.D., Study Director — Incyte Corporation
Locations (19):
- United States (19):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - UC Davis comprehensive Cancer Center, Sacramento, California
  - UCLA Medical Hematology & Oncology, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oncology Hematology Care Clinical Trials LLC, Cincinnati, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - Texas Oncology, Tyler, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Patel MR, Donnellan W, Byrne M, Asch AS, Zeidan AM, Baer MR, Fathi AT, Kuykendall AT, Zheng F, Walker C, Cheng L, Marando C, Savona MR. Phase 1/2 Study of the Pan-PIM Kinase Inhibitor INCB053914 Alone or in Combination With Standard-of-Care Agents in Patients With Advanced Hematologic Malignancies. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):674-686. doi: 10.1016/j.clml.2023.05.002. Epub 2023 May 15. PMID 37290996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 18 US centers and consisted of 4 parts: Parts 1 and 2 evaluated INCB053914 as a monotherapy, and Parts 3 and 4 evaluated INCB053914 as part of a combination therapy with select standard-of-care agents (cytarabine, azacitidine, and ruxolitinib) in participants with advanced malignancies. Note:The study was terminated early based on strategic business decisions and not due to concerns with the safety and tolerability of INCB053914.
Pre-assignment Details: A total of 58 participants were enrolled and treated in Parts 1 and 2 combined and were included in the safety population and the full analysis set.
  A total of 39 participants enrolled and treated in Parts 3 and 4 combined were included in the safety population and the full analysis set.
Groups:
- Parts 1 and 2: INCB053914 100 mg QD: INCB053914 was self-administered orally once a day as a 100mg immediate release monotherapy dose.
- Parts 1 and 2: INCB053914 50 mg BID: INCB053914 was self-administered orally twice day as a 50mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 65 mg BID: INCB053914 was self-administered orally twice day as a 65mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 80 mg BID: INCB053914 was self-administered orally twice day as a 80mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 100 mg BID: INCB053914 was self-administered orally twice day as a 100mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 115 mg BID: INCB053914 was self-administered orally twice day as a 115mg immediate release monotherapy dose.
- Parts 3 and 4: INCB053914 50 mg BID + Cytarabine: Combination Treatment Group A: 50 mg twice a day + I-DAC (intermediate dose cytarabine) was administered at a dose of 1 g/m2 as an infusion as a combination therapy with INCB053914.
- Parts 3 and 4: INCB053914 50 mg BID + Azacitidine: Combination Treatment Group B: INCB053914 50 mg twice a day + Azacitidine was administered at a dose of 75 mg/m2 subcutaneously or via IV per day, as a combination therapy with INCB053914.
- Part 3 and 4 - INCB053914 80 mg BID + Azacitidine: Combination Treatment Group B: INCB053914 80 mg BID + Azacitidine was administered at a dose of 75 mg/m2 subcutaneously or via IV per day, as a combination therapy with INCB053914.
- Part 3 and 4: INCB053914 50 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 50 mg + Ruxolitinib was administered as an oral dose between 5 mg to 25 mg twice per day, as a combination therapy with INCB053914.
- Part 3 and 4: INCB053914 80 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 80 mg BID + Ruxolitinib was administered as an oral dose between 5 mg to 25 mg twice per day, as a combination therapy with INCB053914.
Period: Overall Study
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID | Parts 3 and 4: INCB053914 50 mg BID + Cytarabine | Parts 3 and 4: INCB053914 50 mg BID + Azacitidine | Part 3 and 4 - INCB053914 80 mg BID + Azacitidine | Part 3 and 4: INCB053914 50 mg BID + Ruxolitinib | Part 3 and 4: INCB053914 80 mg BID + Ruxolitinib
Started | 4 | 11 | 4 | 21 | 12 | 6 | 6 | 7 | 9 | 3 | 14
Completed (All participants in each arm discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.) | 0 (All participants discontinued study treatment and withdrew from the study.)
Not Completed | 4 | 11 | 4 | 21 | 12 | 6 | 6 | 7 | 9 | 3 | 14
Not completed — Death | 4 | 8 | 4 | 16 | 9 | 4 | 6 | 7 | 9 | 1 | 3
Not completed — Study Terminated by the Sponsor | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 6
Not completed — Reason for study withdrawal not specified | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Parts 1 and 2: INCB053914 100 mg QD: INCB053914 will be self-administered orally once a day as a 100mg immediate release monotherapy dose.
- Parts 1 and 2: INCB053914 50 mg BID: INCB053914 will be self-administered orally twice day as a 50mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 65 mg BID: INCB053914 will be self-administered orally twice day as a 65mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 80 mg BID: INCB053914 will be self-administered orally twice day as a 80mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 100 mg BID: INCB053914 will be self-administered orally twice day s a 100mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 115 mg BID: INCB053914 will be self-administered orally twice day as a 115mg immediate release monotherapy dose.
- Parts 3 and 4: INCB053914 50 mg BID + Cytarabine: Combination Treatment Group A: 50 mg BID + I-DAC (intermediate dose cytarabine) will be administered at a dose of 1 g/m2 per day as an infusion as a combination therapy with INCB053914.
- Parts 3 and 4: INCB053914 50 mg BID + Azacitidine: Combination Treatment Group B: Azacitidine will be administered at a dose of 75 mg/m2 subcutaneously or via IV per day, as a combination therapy with INCB053914 50 mg BID.
- Part 3 and 4 - INCB053914 80 mg BID + Azacitidine: Combination Treatment Group B: INCB053914 80 mg BID + Azacitidine will be administered at a dose of 75 mg/m2 subcutaneously or via IV per day, as a combination therapy with INCB053914.
- Part 3 and 4: INCB053914 50 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 50 mg BID + Ruxolitinib will be administered as an oral dose between 5 mg to 25 mg twice per day, as a combination therapy with INCB053914.
- Part 3 and 4: INCB053914 80 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 80 mg + Ruxolitinib will be administered as an oral dose between 5 mg to 25 mg twice per day, as a combination therapy with INCB053914.
- Total: Total of all reporting groups
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID | Parts 3 and 4: INCB053914 50 mg BID + Cytarabine | Parts 3 and 4: INCB053914 50 mg BID + Azacitidine | Part 3 and 4 - INCB053914 80 mg BID + Azacitidine | Part 3 and 4: INCB053914 50 mg BID + Ruxolitinib | Part 3 and 4: INCB053914 80 mg BID + Ruxolitinib | Total
Number analyzed (Participants) | 4 | 11 | 4 | 21 | 12 | 6 | 6 | 7 | 9 | 3 | 14 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (14.25) | 67.1 (14.64) | 67.3 (9.18) | 70.8 (11.50) | 76.5 (7.19) | 70.5 (9.67) | 70.8 (6.46) | 60.9 (20.83) | 72.9 (6.31) | 70.0 (5.0) | 72.6 (7.48) | 70.2 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 11 | 3 | 3 | 5 | 5 | 2 | 2 | 6 | 47
  Male | 1 | 6 | 2 | 10 | 9 | 3 | 1 | 2 | 7 | 1 | 8 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 4 | 11 | 1 | 16 | 11 | 5 | 4 | 7 | 8 | 3 | 13 | 83
  Black/African American | 0 | 0 | 3 | 4 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 11
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 3 | 11 | 4 | 18 | 12 | 6 | 6 | 7 | 8 | 3 | 11 | 89
  Unknown | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Safety and Tolerability of INCB053914 as Measured by the Number of Participants With Adverse Events
Time Frame: Approximately 7 months
Measure: Number; unit: Participants
Groups:
- Parts 1 and 2: INB053914 65 mg BID: INCB053914 will be self-administered orally twice day in as a 65mg immediate release monotherapy dose
- Parts 1 and 2: INB053914 80 mg BID: INCB053914 will be self-administered orally twice day in as a 80mg immediate release monotherapy dose.
- Parts 1 and 2: INB053914 100 mg BID: INCB053914 will be self-administered orally twice day as a 100mg immediate release monotherapy dose.
- Parts 3 and 4: INCB053914 50 mg BID + Cytarabine: Combination Treatment Group A: INCB053914 50 mg BID + Cytarabine
- Parts 3 and 4: INCB053914 50 mg BID + Azacitidine: Combination Treatment Group B: INCB053914 50 mg BID + Azacitidine
- Parts 3 and 4: INCB053914 80 mg BID + Azacitine: Combination Treatment Group B: INCB053914 80 mg BID + Azacitine
- Parts 3 & 4: INCB 053914 50 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 50 mg BID + Ruxolitinib
- Parts 3 & 4: INCB 053914 80 mg + Ruxolitinib: Combination Treatment Group C: INCB 053914 80 mg BID + Ruxolitinib
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID | Parts 3 and 4: INCB053914 50 mg BID + Cytarabine | Parts 3 and 4: INCB053914 50 mg BID + Azacitidine | Parts 3 and 4: INCB053914 80 mg BID + Azacitine | Parts 3 & 4: INCB 053914 50 mg BID + Ruxolitinib | Parts 3 & 4: INCB 053914 80 mg + Ruxolitinib
Number analyzed (Participants) | 4 | 11 | 4 | 21 | 12 | 3 | 6 | 7 | 9 | 3 | 14
Participants | 4 | 11 | 4 | 21 | 12 | 6 | 6 | 7 | 9 | 3 | 14

2. Primary Outcome: Part 4 Only : Determination of the Efficacy of INCB053914 in Combination With the Intermediate-dose Cytarabine (I DAC) in Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML) Based on Objective Remission Rate (ORR)
Description: The primary efficacy endpoint of ORR in patients with AML who received INCB053914 in combination with cytarabine in Part 4 was not assessed because Part 4 was not opened for enrollment owing to this combination regimen not being tolerated in Part 3.
Time Frame: Approximately 2 months
Population: Part 4 was not opened for enrollment owing to combination regimen not being tolerated in Part 3.
Groups:
- Part 4: INCB053914 50 mg BID + Cytarabine): Combination Treatment Group A: INCB053914 50 mg BID + Cytarabine
Arm/Group | Part 4: INCB053914 50 mg BID + Cytarabine)
Number analyzed (Participants) | 0

3. Primary Outcome: Part 4 Only : Determination of the Efficacy of INCB053914 in Combination With Azacitidine in Subjects With Newly Diagnosed AML Who Are 65 Years or Older and Unfit for Intensive Chemotherapy Based on ORR
Description: The primary efficacy endpoint of ORR in patients with AML who received INCB053914 plus azacitidine in Part 4 was not performed due to limited enrollment as a result of early study termination.
Time Frame: Approximately 6 months
Population: Part 4 was not opened for enrollment.
Groups:
- Part 4: INCB053914 50 mg BID + Azacitidine: Combination Treatment Group B INCB053914 50 mg BID + Azacitidine
- Part 4: INB053914 80 mg BID + Azactidine: Combination Treatment Group B: B053914 80 mg BID + Azactidine
Arm/Group | Part 4: INCB053914 50 mg BID + Azacitidine | Part 4: INB053914 80 mg BID + Azactidine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Evaluation of Phosphorylated BCL--2 Associated Death Promoter Protein (pBAD)
Description: Percent Inhibition of pBAD at the C1D15 trough from the pBAD at pre-dose by ex vivo cellular assay
Time Frame: 1 month
Population: The PD evaluable population includes those in the safety population who have at least 1 valid PD measurements at both pre- and postdose.
Measure: Mean (Full Range); unit: Percentage of Inhibition
Groups:
- Parts 1 and 2: INCB053914 50 mg BID: INCB053914 will be self-administered orally twice day in as a 50mg immediate release tablet as a monotherapy.
- Parts 1 and 2: INB053914 65 mg BID: INCB053914 will be self-administered orally twice day in as a 65mg immediate release tablet as a monotherapy.
- Parts 1 and 2: INB053914 80 mg BID: INCB053914 will be self-administered orally twice day in as a 80mg immediate release tablet as a monotherapy.
- Parts 1 and 2: INB053914 115 mg BID: INCB053914 will be self-administered orally twice day in as a 115mg immediate release tablet as a monotherapy.
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 4 | 10 | 3 | 3 | 8 | 3
Percentage of Inhibition | 41 [16 to 67] | 37 [17 to 59] | 68 [52 to 91] | 78 [63 to 104] | 55 [28 to 92] | 58 [34 to 80]

5. Secondary Outcome: Pharmacokinetics: Tmax of Combination Treatment Group A INCB053914 50 mg + Cytarabine
Time Frame: Cycle 1 Day 5
Measure: Median (Full Range); unit: h
Groups:
- Parts 3 & 4: INCB053914 50 mg BID + Cytarabine: Combination Group A: INCB053914 50 mg BID + Cytarabine
Arm/Group | Parts 3 & 4: INCB053914 50 mg BID + Cytarabine
Number analyzed (Participants) | 6
h | 1.52 [1 to 2.07]

6. Secondary Outcome: Pharmacokinetics: AUCtau of Combination Treatment Group A INCB053914 50 mg + Cytarabine
Time Frame: Cycle 1 Day 5
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Parts 3 & 4: INCB053914 50 mg BID + Cytarabine
Number analyzed (Participants) | 6
nM*h | 2860 (2040)

7. Secondary Outcome: Pharmacokinetics: Cl/F of Combination Treatment Group A INCB053914 50 mg + Cytarabine
Time Frame: Cycle 1 Day 5
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Parts 3 & 4: INCB053914 50 mg BID + Cytarabine
Number analyzed (Participants) | 6
L/hr | 122 (213)

8. Secondary Outcome: Pharmacokinetics: Cmax of Combination Treatment Group A INCB053914 50 mg + Cytarabine
Time Frame: Cycle 1 Day 5
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INCB053914 50 mg BID + Cytarabine
Number analyzed (Participants) | 6
nM | 423 (283)

9. Secondary Outcome: Pharmacokinetics: Cmin of Combination Treatment Group A INCB053914 50 mg + Cytarabine
Time Frame: Cycle 1 Day 5
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INCB053914 50 mg BID + Cytarabine
Number analyzed (Participants) | 6
nM | 139 (101)

10. Secondary Outcome: Pharmacokinetics: Tmax of Combination Group B INCB053914 80 mg + Azatcitidine
Time Frame: Cycle 1 Day 8
Measure: Median (Full Range); unit: h
Groups:
- Parts 3 & 4: INCB053914 80 mg BID + Azacitidine: Combination Treatment Group B: INCB053914 80 mg BID + Azacitidine
Arm/Group | Parts 3 & 4: INCB053914 80 mg BID + Azacitidine
Number analyzed (Participants) | 7
h | 2 [1 to 4]

11. Secondary Outcome: Pharmacokinetics: AUCtau of Combination Group B INCB053914 80 mg + Azatcitidine
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Parts 3 & 4: INCB053914 80 mg BID + Azacitidine
Number analyzed (Participants) | 7
nM*h | 11000 (11100)

12. Secondary Outcome: Pharmacokinetics: Cl/F of Combination Group B INCB053914 80 mg + Azatcitidine
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Parts 3 & 4: INCB053914 80 mg BID + Azacitidine
Number analyzed (Participants) | 7
L/h | 30.8 (24.7)

13. Secondary Outcome: Pharmacokinetics: Cmax of Combination Group B INCB053914 80 mg + Azatcitidine
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INCB053914 80 mg BID + Azacitidine
Number analyzed (Participants) | 7
nM | 1320 (1240)

14. Secondary Outcome: Pharmacokinetics: Cmin of Combination Group B INCB053914 80 mg + Azatcitidine
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INCB053914 80 mg BID + Azacitidine
Number analyzed (Participants) | 7
nM | 513 (431)

15. Secondary Outcome: Pharmacokinetics: Tmax of Combination Treatment Group C INCB053914 80 mg + Ruxolitinib
Time Frame: Regimen 2 Week 4
Measure: Median (Full Range); unit: h
Groups:
- Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib: Combination Treatment Group C: INCB053914 80 mg BID + Ruxolitinib
Arm/Group | Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib
Number analyzed (Participants) | 6
h | 2.02 [1 to 4]

16. Secondary Outcome: Pharmacokinetics: AUCtau of Combination Treatment Group C INCB053914 80 mg + Ruxolitinib
Time Frame: Regimen 2 Week 4
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib
Number analyzed (Participants) | 6
nM*h | 3060 (1730)

17. Secondary Outcome: Pharmacokinetics: Cl/F of Combination Treatment Group C INCB053914 80 mg + Ruxolitinib
Time Frame: Regimen 2 Week 4
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib
Number analyzed (Participants) | 6
L/h | 69.7 (41.1)

18. Secondary Outcome: Pharmacokinetics: Cmax of Combination Treatment Group C INCB053914 80 mg + Ruxolitinib
Time Frame: Regimen 2 Week 4
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib
Number analyzed (Participants) | 6
nM | 541 (376)

19. Secondary Outcome: Pharmacokinetics: Cmin of Combination Treatment Group C INCB053914 80 mg + Ruxolitinib
Time Frame: Regimen 2 Week 4
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 3 & 4: INB053914 80 mg BID + Ruxolitinib
Number analyzed (Participants) | 6
nM | 104 (63.7)

20. Secondary Outcome: Pharmacokinetics: Tmax of INCB053914 Monotherapy
Time Frame: Cycle 1 Day 8
Measure: Median (Full Range); unit: hour
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 3 | 8 | 3 | 14 | 11 | 2
hour | 2.0 [1.0 to 2.2] | 1.0 [0.5 to 4.0] | 2.0 [2.0 to 4.0] | 1.5 [0.5 to 4.1] | 1.0 [.5 to 2.2] | NA [1.0 to 1.1] — Individual values presented given N=2

21. Secondary Outcome: Pharmacokinetics: AUCtau of INCB053914 Monotherapy
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 3 | 8 | 3 | 14 | 11 | 2
nM*h | 4140 (282) | 1290 (924) | 2480 (2470) | 3940 (3120) | 5410 (5060) | 5630 (764)

22. Secondary Outcome: Pharmacokinetics: CL/F of INCB053914 Monotherapy
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 3 | 8 | 3 | 14 | 11 | 2
L/h | 47.2 (3.16) | 132 (132) | 95.1 (73.2) | 71.2 (58.5) | 85.2 (114) | 39.8 (293)

23. Secondary Outcome: Pharmacokinetics: Cmax of INCB053914 Monotherapy
Time Frame: Cycle 1 Day 8
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 3 | 8 | 3 | 14 | 11 | 2
nM | 352 (126) | 227 (188) | 333 (276) | 591 (447) | 796 (659) | 578 (131)

24. Secondary Outcome: Pharmacokinetics: Ctau of INCB053914 Monotherapy
Time Frame: Cycle 1 Day 8
Population: Ctau was calculated using the predose value on C1D8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Parts 1 and 2: INCB053914 100 mg QD | Parts 1 and 2: INCB053914 50 mg BID | Parts 1 and 2: INB053914 65 mg BID | Parts 1 and 2: INB053914 80 mg BID | Parts 1 and 2: INB053914 100 mg BID | Parts 1 and 2: INB053914 115 mg BID
Number analyzed (Participants) | 3 | 9 | 3 | 14 | 11 | 5
L/h | 98.2 (44.9) | 65.7 (44.2) | 132 (148) | 213 (188) | 293 (322) | 410 (482)

ADVERSE EVENTS:
Time Frame: up to approximately 6 months
Groups:
- Part 1 and 2 - INCB053914: 100 mg QD: Part 1 and 2 - INCB053914: 100 mg QD
- Part 1 and 2 - INCB053914: 50 mg BID: Part 1 and 2 - INCB053914: 50 mg BID
- Part 1 and 2 - INCB053914: 65 mg BID: Part 1 and 2 - INCB053914: 65 mg BID
- Part 1 and 2 - INCB053914: 80 mg BID: Part 1 and 2 - INCB053914: 80 mg BID
- Part 1 and 2 - INCB053914: 100 mg BID: Part 1 and 2 - INCB053914: 100 mg BID
- Part 1 and 2 - INCB053914: 115 mg BID: Part 1 and 2 - INCB053914: 115 mg BID
- Part 3 and 4 - INCB053914: 50 mg BID + Cytarabine: Part 3 and 4 - INCB053914: 50 mg BID + Cytarabine
- Part 3 and 4 - INCB053914: 50 mg BID + Azacitidine: Part 3 and 4 - INCB053914: 50 mg BID + Azacitidine
- Part 3 and 4 - INCB053914: 80 mg BID + Azacitidine: Part 3 and 4 - INCB053914: 80 mg BID + Azacitidine
- Part 3 and 4 - INCB053914: 50 mg BID + Ruxolitinib: Part 3 and 4 - INCB053914: 50 mg BID + Ruxolitinib
- Part 3 and 4 - INCB053914: 80 mg BID + Ruxolitinib: Part 3 and 4 - INCB053914: 80 mg BID + Ruxolitinib
Arm/Group | Part 1 and 2 - INCB053914: 100 mg QD | Part 1 and 2 - INCB053914: 50 mg BID | Part 1 and 2 - INCB053914: 65 mg BID | Part 1 and 2 - INCB053914: 80 mg BID | Part 1 and 2 - INCB053914: 100 mg BID | Part 1 and 2 - INCB053914: 115 mg BID | Part 3 and 4 - INCB053914: 50 mg BID + Cytarabine | Part 3 and 4 - INCB053914: 50 mg BID + Azacitidine | Part 3 and 4 - INCB053914: 80 mg BID + Azacitidine | Part 3 and 4 - INCB053914: 50 mg BID + Ruxolitinib | Part 3 and 4 - INCB053914: 80 mg BID + Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 4/4 | 8/11 | 4/4 | 19/21 | 9/12 | 4/6 | 6/6 | 7/7 | 9/9 | 1/3 | 3/14
Serious Adverse Events (participants affected / at risk) | 3/4 | 6/11 | 3/4 | 6/21 | 8/12 | 5/6 | 5/6 | 5/7 | 6/9 | 0/3 | 5/14
Other Adverse Events (participants affected / at risk) | 4/4 | 11/11 | 4/4 | 20/21 | 12/12 | 6/6 | 6/6 | 7/7 | 8/9 | 3/3 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 and 2 - INCB053914: 100 mg QD (N=4) | Part 1 and 2 - INCB053914: 50 mg BID (N=11) | Part 1 and 2 - INCB053914: 65 mg BID (N=4) | Part 1 and 2 - INCB053914: 80 mg BID (N=21) | Part 1 and 2 - INCB053914: 100 mg BID (N=12) | Part 1 and 2 - INCB053914: 115 mg BID (N=6) | Part 3 and 4 - INCB053914: 50 mg BID + Cytarabine (N=6) | Part 3 and 4 - INCB053914: 50 mg BID + Azacitidine (N=7) | Part 3 and 4 - INCB053914: 80 mg BID + Azacitidine (N=9) | Part 3 and 4 - INCB053914: 50 mg BID + Ruxolitinib (N=3) | Part 3 and 4 - INCB053914: 80 mg BID + Ruxolitinib (N=14)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 and 2 - INCB053914: 100 mg QD (N=4) | Part 1 and 2 - INCB053914: 50 mg BID (N=11) | Part 1 and 2 - INCB053914: 65 mg BID (N=4) | Part 1 and 2 - INCB053914: 80 mg BID (N=21) | Part 1 and 2 - INCB053914: 100 mg BID (N=12) | Part 1 and 2 - INCB053914: 115 mg BID (N=6) | Part 3 and 4 - INCB053914: 50 mg BID + Cytarabine (N=6) | Part 3 and 4 - INCB053914: 50 mg BID + Azacitidine (N=7) | Part 3 and 4 - INCB053914: 80 mg BID + Azacitidine (N=9) | Part 3 and 4 - INCB053914: 50 mg BID + Ruxolitinib (N=3) | Part 3 and 4 - INCB053914: 80 mg BID + Ruxolitinib (N=14)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (2) | 8 (10) | 4 (5) | 2 (2) | 4 (4) | 1 (1) | 4 (8) | 0 (0) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 3 (4) | 5 (10) | 5 (22) | 2 (2) | 3 (9) | 3 (4) | 3 (3) | 1 (4) | 5 (9)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (3) | 1 (2) | 7 (9) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 4 (6) | 0 (0) | 6 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 4 (4) | 3 (4) | 3 (4) | 4 (5) | 3 (5) | 3 (5) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 4 (4) | 1 (1) | 5 (6) | 6 (6) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (9) | 0 (0) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 1 (2) | 2 (3) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (6) | 1 (1) | 4 (4) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (7) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (7) | 0 (0) | 5 (9)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 3 (4)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT02587598/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02587598/SAP_001.pdf